CLINICAL TRIAL: NCT05690646
Title: Prophylactic Effect of Nirmatrelvir/Ritonavir and Ursodeoxycholic Acid on Reducing Complications After Cardiac Surgery During COVID-19 Pandemics: A Prospective, Randomized Controlled, Multicenter Trial
Brief Title: Prophylactic Effect of Nirmatrelvir/Ritonavir and Ursodeoxycholic Acid on Reducing Complications After Cardiac Surgery
Acronym: PEP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCRC2023001
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — nirmatrelvir and ritonavir drug combination; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NR group (Experimental): nirmatrelvir 300mg q12h and ritonavir 100 mg q12h for 5 days
  Interventions: Drug: Nirmatrelvir/ritonavir
- UA group (Experimental): ursodeoxycholic acid group, 15mg/kg/day bid for5 days
  Interventions: Drug: Ursodeoxycholic acid
- combination group (Experimental): nirmatrelvir 300mg q12h and ritonavir 100 mg q12h for 5 days and ursodeoxycholic acid group, 15mg/kg/day bid for5 days
  Interventions: Drug: Nirmatrelvir/ritonavir; Drug: Ursodeoxycholic acid
- control group (No Intervention): No intervention

INTERVENTIONS:
Drug: Nirmatrelvir/ritonavir — nirmatrelvir 300mg q12h and ritonavir 100 mg q12h for 5 days
  Arms: NR group; combination group
Drug: Ursodeoxycholic acid — ursodeoxycholic acid 15mg/kg/day bid for5 days
  Arms: UA group; combination group

SUMMARY:
Prophylactic effect of nirmatrelvir/ritonavir and ursodeoxycholic acid on reducing complications after cardiac surgery during covid-19 pandemics (the pep trial) is a multicenter, randomized controlled trial. The aim of the pep trial is to investigate whether prophylactic use of nirmatrelvir/ritonavir and ursodeoxycholic could reduce complications after cardiac surgery.

DETAILED DESCRIPTION:
After informed consent, four centers and 436 eligible admissions will be recruited. Eligible patients would be randomized (1:1:1:1) to nirmatrelvir/ritonavir group (nirmatrelvir 300mg q12h and ritonavir 100 mg q12h for 5 days), ursodeoxycholic acid group (ursodeoxycholic acid group, 15mg/kg/day bid for5 days), combination group (nirmatrelvir/ritonavir and ursodeoxycholic acid for 5days) and control group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* COVID-19 nucleic acid test or antigen test positive history, without symptom or recover from COVID-19 related symptoms ≥2 weeks
* Receive open-chest cardiac surgery
* COVID-19 nucleic acid test and antigen test negative and no signs of pneumonia in chest CT
* Patients with written informed consent.

Exclusion Criteria:

* Emergency surgery
* eGFR ≤30ml/min
* Severe liver dysfunction
* Contraindication to nirmatrelvir/ritonavir or ursodeoxycholic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
MACCE | 30 days after surgery or during hospitalization
  All-cause mortality, myocardial infarction, stroke, moderate to severe acute kidney injury, and COVID-19 pneumonia

SECONDARY OUTCOMES:
All-cause mortality | 30 days after surgery or during hospitalization
  All-cause mortality
Rate of Myocardial infarction | 30 days after surgery or during hospitalization
  new onset of myocardial infarction
Rate of Stroke | 30 days after surgery or during hospitalization
  new onset of stroke
Rate of Moderate to severe acute kidney injury | 30 days after surgery or during hospitalization
  new onset of moderate to severe acute kidney injury
Rate of COVID-19 pneumonia | 30 days after surgery or during hospitalization
  new onset of COVID-19 pneumonia
Rate of Cardiogenic death | 30 days after surgery or during hospitalization
  Cardiogenic death
Rate of Severe pneumonia | 30 days after surgery or during hospitalization
  new onset of Severe pneumonia
Rate of Ventilation ≥24h | 30 days after surgery or during hospitalization
  Ventilation ≥24h after surgery
Rate of Pulmonary embolism | 30 days after surgery or during hospitalization
  new onset of Pulmonary embolism
Rate of Re-operation for bleeding | 30 days after surgery or during hospitalization
  Re-operation for bleeding after primary surgery
All-cause mortality | 1 year after surgery
  All-cause mortality
Rate of Myocardial infarction | 1 year after surgery
  new onset of Myocardial infarction
Rate of Stroke | 1 year after surgery
  new onset of Stroke
Rate of Renal insufficiency | 1 year after surgery
  new onset of Renal insufficiency
Rate of Re-hospitalization for respiratory disease | 1 year after surgery
  Re-hospitalization for respiratory disease
Rate of Cardiogenic re-hospitalization | 1 year after surgery
  Cardiogenic re-hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No